CLINICAL TRIAL: NCT01382121
Title: Increasing Self-efficacy and VO2 Max Scores in Obese Adolescents: a Peer Modeling Intervention
Brief Title: Adolescent Fitness Assessment Program
Acronym: AFAP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PeakVO2 PM RCT
Record Dates: First submitted 2011-04-21; First posted 2011-06-27 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes
Keywords: Peer modeling; Observational learning; Obesity; Adolescents; Maximum ventilatory oxygen; Aerobic fitness; Health behaviour
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer modeling (Experimental): Participants watch a video geared to increase confidence in ability to preform fitness test. Male participants will watch a video of a male adolescent completing the fitness test and talking about coping mechanisms used to preform to the best of his ability. Female participants will watch a video of a female adolescent completing the fitness test and talking about coping mechanisms used to preform to the best of her ability.
  Interventions: Behavioral: Peer Modeling
- Control (Active Comparator): Participants watch a video unrelated to the fitness test and self-efficacy. The video depicts healthy food and nutrition options.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Peer Modeling — Participants watch a video of an adolescent completing the fitness test and explaining coping mechanisms to preform the test well.
  Other Names: Observational Learning; Coping Model
  Arms: Peer modeling
Behavioral: Control — watching a video unrelated to the fitness test and self-efficacy
  Other Names: Contact control; Active control
  Arms: Control

SUMMARY:
The purpose of this study is to implement a peer modeling intervention to improve self-efficacy and aerobic fitness in obese youth. A total of 40 obese (defined as Body Mass Index greater than the 95th percentile for age and gender) youth will participate in this study.

DETAILED DESCRIPTION:
There has been a dramatic increase in the prevalence of overweight and obese children in all regions of Canada. In fact, Canada has one of the highest rates of childhood obesity compared to other developed countries. This is disconcerting because this preventative condition is strongly associated with the risk of future disease, such as adult obesity, insulin resistance, type 2 diabetes, cardiovascular problems and psychosocial distress. This trend is a driving factor to develop effective strategies for assessment and intervention.

Aerobic fitness is the ability of the cardiovascular and respiratory system to deliver oxygen to working muscles and utilize that oxygen to produce energy. Aerobic fitness is a strong indicator of physical activity and also correlates with the aforementioned diseases. It is measured as peak ventilatory oxygen (peak VO2; mL/kg min), and is evaluated using a maximal incremental exercise protocol on a treadmill, whereby expired gases are analyzed using a metabolic cart. Aerobic fitness values are inconsistent in youth, particularly obese youth. This discrepancy is due to low self-efficacy. Self-efficacy refers to the belief that one has the power and capabilities to produce an effect. Low self-efficacy is prominent in obese youth because they lack actual and perceived physical competence and social support. This may translate into less effort invested by this population into physical activity, and by the same token, aerobic fitness tests. To date, no experimental studies have attempted to address these psychological variables and apply an intervention to achieve accurate peak VO2 values in obese adolescents.

Peer modelling is the demonstration of particular behaviors that are learned observationally and is a powerful source of self-efficacy. This mode of learning has been very successful in increasing the consumption of new foods (36 subjects) and activity levels (100 subjects) in children. Based on this success, it would suggest that the investigators could confidently apply it to this study. Therefore the main objective is to examine the effect of a modeling intervention (DVD film) on self-efficacy and peak VO2 in obese youth during a maximal treadmill test. Models will demonstrate and articulate increased confidence to perform the test and offer a variety of strategies to cope with the maximal effort and overcome the associated challenges during the test (e.g. shortness of breath, sweating, and increased heart rate). The models will not be participants in the study.

Obese (defined as Body Mass Index greater than the 95th percentile for age and gender) youth (10-17 years, N = 40) who receive written consent from a parent or guardian will be asked to participate in the study. Prior to undertaking the aerobic fitness test, children are required to seek approval from their family physician by completing the Physical Activity Readiness Questionnaire (PAR-Q).

Participants will be randomized after baseline measures are completed into one of two conditions: peer modeling intervention or control to ensure group equivalency. Following randomization, participants in the intervention group will watch the peer modeling DVD film in the lab. Those in the control group will view a DVD film of similar length about nutrition. After seven days, participants in both groups will return for follow-up. One week is a suitable interval because it provides time for participants to reflect on any information they received from the DVD films and minimize external confounding factors, while not providing enough time to see changes in fitness (which requires approximately 3 months). Prior to the second exercise test, participants will watch the DVD film they viewed the previous week. Afterwards, participants will complete their peak VO2 test and self-reported measures. All participants will be asked not to change their normal physical activity patterns during the week.

To complete a peak VO2 test, participants will be required to complete a maximal incremental exercise protocol on a treadmill. The test will be conducted by trained personnel and terminated when participants are unable to continue the protocol, or when their vital signs warranted discontinuation.

The results of this RCT will provide an accurate measurement of aerobic fitness, which is crucial to assessing health status, risk of disease and assisting in planning programs aimed at improving quality of life in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 10-17 years who are obese, defined as Body Mass Index greater than the 95th percentile for age and gender

Exclusion Criteria:

* Participants who smoke, are pregnant or have an illness or disease will be excluded from the study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Physiological measure: Aerobic Fitness | Baseline (day 1) and follow-up (day 7)
  Changes in aerobic fitness from baseline (day 1) to follow-up (day 7) will be evaluated by a trained exercise physiologist using a standardized, maximal incremental exercise protocol (Modified Bruce protocol) on a treadmill. Expired gases will be analyzed using a metabolic cart (Cosmed Quark B2 cardiopulmonary testing, Image Monitoring). Peak oxygen consumption (Peak VO2) will be determined by taking the highest values during a 15 second period and expressed in absolute (l/min) and relative (ml/kg/min) units with the latter unit used for subsequent analysis.
Psychological: Self-Efficacy | Baseline (day 1) and follow-up (day 7)
  Changes in self-efficacy from baseline (day 1) to follow-up (day 7) will be evaluated by an 18-item Self-Efficacy Scale (adapted from McAuley & Milhalko, 1998) to evaluate participants' confidence to successfully perform increasing intensities and durations of physical activity.

SECONDARY OUTCOMES:
Changes in variability (standard deviation) | Baseline (day 1) and follow-up (day 7)
  Changes in variability (standard deviation) in the aerobic fitness and self-efficacy data will be analyzed using statistical software.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, PhD, Principal Investigator — The University of Western Ontario
Locations (1):
- Exercise and Health Psychology Laboratory, London, Ontario, Canada

REFERENCES:
- [Background] Willms JD, Tremblay MS, Katzmarzyk PT. Geographic and demographic variation in the prevalence of overweight Canadian children. Obes Res. 2003 May;11(5):668-73. doi: 10.1038/oby.2003.95. PMID 12740457
- [Background] Cairney J, Hay JA, Faught BE, Leger L, Mathers B. Generalized self-efficacy and performance on the 20-metre shuttle run in children. Am J Hum Biol. 2008 Mar-Apr;20(2):132-8. doi: 10.1002/ajhb.20690. PMID 17990324
- [Background] Carrel AL, Sledge JS, Ventura SJ, Clark RR, Peterson SE, Eickhoff J, Allen DB. Measuring aerobic cycling power as an assessment of childhood fitness. J Strength Cond Res. 2007 Aug;21(3):685-8. doi: 10.1519/R-22606.1. PMID 17685725
- [Background] Korsten-Reck U, Kaspar T, Korsten K, Kromeyer-Hauschild K, Bos K, Berg A, Dickhuth HH. Motor abilities and aerobic fitness of obese children. Int J Sports Med. 2007 Sep;28(9):762-7. doi: 10.1055/s-2007-964968. Epub 2007 May 11. PMID 17497579
- [Background] Jones RA, Okely AD, Caputi P, Cliff DP. Perceived and actual competence among overweight and non-overweight children. J Sci Med Sport. 2010 Nov;13(6):589-96. doi: 10.1016/j.jsams.2010.04.002. Epub 2010 Jul 2. PMID 20580314
- [Background] Greenhalgh J, Dowey AJ, Horne PJ, Fergus Lowe C, Griffiths JH, Whitaker CJ. Positive- and negative peer modelling effects on young children's consumption of novel blue foods. Appetite. 2009 Jun;52(3):646-653. doi: 10.1016/j.appet.2009.02.016. Epub 2009 Mar 6. PMID 19501762
- [Background] Horne PJ, Hardman CA, Lowe CF, Rowlands AV. Increasing children's physical activity: a peer modelling, rewards and pedometer-based intervention. Eur J Clin Nutr. 2009 Feb;63(2):191-8. doi: 10.1038/sj.ejcn.1602915. Epub 2007 Sep 19. PMID 17882131
- See also: Exercise and Health Psychology Laboratory — http://www.ehpl.uwo.ca